CLINICAL TRIAL: NCT05603988
Title: Evaluation of The Effect of 980nm Diode Laser Intracanal Irradiation on Levels of Interleukin-8 Expression in Lesions Refractory to Endodontic Treatment: A Randomized Control Trial
Brief Title: Evaluation of The Effect of 980nm Diode Laser Intracanal Irradiation on Levels of Interleukin-8 Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Ahmed Morsy, lecturer in endodontic department, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAMorsy
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Endodontically Treated Teeth
Keywords: Diode laser; Endodontic retreatment; IL-8 expression
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): • Mock laser application (Placebo group): The fiber optic tip will be inserted inside the root canal, mimicking the laser irradiation group, but not activated
  Interventions: Other: Placebo
- Diode Laser group (Other): Intracanal Diode laser application
  Interventions: Device: Intracanal Diode laser irradiation

INTERVENTIONS:
Device: Intracanal Diode laser irradiation — After endodontic retreatment, root canals will be irradiated with a 980 nm diode laser coupled with optical fibre 200 μm (Litemedics, Italy) with setting 1.2-watt power, in pulsed mode. The irradiation protocol will be of 5-sec irradiation followed by a 10-sec pause, which constituted one lasing cycle. The lasing cycle will be performed four times for each tooth. The tip will be positioned 1 mm short of the apex. Followed by activation during which it will be slowly dragged at a speed of approximately 2 mm/ sec in a way that the root canals will be irradiated from the apical to the coronal portion, in a helicoidal movement touching the canal walls.
  Arms: Diode Laser group
Other: Placebo — After endodontic retreatment, mock laser application (Placebo group) will be applied:
  The fiberoptic tip will be inserted inside the root canal, mimicking the laser irradiation group, but not activated
  Arms: Placebo group

SUMMARY:
This clinical trial will be conducted to evaluate the amount of Il-8 expression before and after the application of intracanal irradiation with diode laser 980 nm versus placebo in failed endodontic cases with periapical lesions.

DETAILED DESCRIPTION:
* Thorough medical and dental history for the eligible patients
* Thorough intraoral and extraoral diagnosis
* Local anesthesia
* Isolation and removal of any previous filling or restoration
* Removal of old gutta percha and establish patency to the full working length.
* 1st sample: will be collected using 3 sterile paper points
* Chemo-mechanical preparation.
* 2nd sample collection

  • Laser group: The canals will be irradiated with a high-power diode laser, with wavelength of 980 nm, maximum output of 3 watts and coupled with a fiber optic tip of 200 µm diameter.

  • Mock laser application (Placebo group): The fiberoptic tip will be inserted inside the root canal, mimicking the laser irradiation, but not activated.
* 3rd sample collection
* A piece of dry cotton will be placed in the access cavity, and then will be sealed with glass ionomer filling material
* 2nd visit: 1 week later, 4th sample collection then Obturation
* Number of visits & follow up period: Two visits

ELIGIBILITY:
Inclusion Criteria:

* failed previously treated endodontic single-rooted teeth with chronic periapical lesions; with radiographic evidence of periapical radiolucency of not less than 1 cm diameter will be selected.
* Teeth with straight root canals.
* No contributory medical history.
* No previous administration of analgesics and/or antibiotics within the previous 2 weeks.

Exclusion Criteria:

* Retreatment cases with complications such as separated instruments, perforations, ledges, resorption, transportation, calcifications, immature apices and over fillings.
* Teeth with curved roots.
* Swelling or sinus tract.
* Mutilated teeth that interfere with proper isolation and seal between visits.
* Subjects with generalized periodontitis, or if the tooth has a probing depth of more than 3 mm.
* Subjects with uncontrolled diabetes or debilitating diseases.
* Pregnant or nursing females.
* Systemic disorders that necessitate antibiotic prophylaxis or prevent the use of Ibuprofen.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
quantification of IL-8 | one week
  - After collection of all the samples, quantification of IL-8 will be determined using ELISA kit before (S-1), after chemo-mechanical preparation (S-2), after intracanal irradiation or placebo effect (S-3) and last after one week of the treatment (S-4). The kit is used according to the manufacturer's recommendations.

SECONDARY OUTCOMES:
Postoperative pain | 6, 12, 24 hours and 7 days
  Following the first visit, the modified visual analogue scale (VAS scale) with 11 points where 0 means no pain and 10 means maximum pain will be used to record patient's level of pain

CONTACTS AND LOCATIONS:
Overall Officials: Dina A Morsy, lecturer, Principal Investigator — Cairo University; Sherif A Elkhodary, assoc. Prof, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morsy DA, Negm M, Diab A, Ahmed G. Postoperative pain and antibacterial effect of 980 nm diode laser versus conventional endodontic treatment in necrotic teeth with chronic periapical lesions: A randomized control trial. F1000Res. 2018 Nov 15;7:1795. doi: 10.12688/f1000research.16794.1. eCollection 2018. PMID 31372210
- [Result] Kamma JJ, Vasdekis VG, Romanos GE. The effect of diode laser (980 nm) treatment on aggressive periodontitis: evaluation of microbial and clinical parameters. Photomed Laser Surg. 2009 Feb;27(1):11-9. doi: 10.1089/pho.2007.2233. PMID 19196111